CLINICAL TRIAL: NCT00006318
Title: Role of Prostaglandins in the Control of Cerebral Blood Flow During Hypercapnia and Functional Activation in Humans
Brief Title: Role of Prostaglandins in the Regulation of Brain Blood Flow
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000226; 00-CC-0226
Record Dates: First submitted 2000-09-30; First posted 2000-10-02 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-12

CONDITIONS: Healthy; Hypercapnia
Keywords: Cerebral Blood Flow; CO2 Inhalation; Imaging; MRI; Perfusion; Functional Activation
MeSH Terms: conditions — Hypercapnia

SUMMARY:
This study will use magnetic resonance imaging (MRI) to examine the role of prostaglandins-a type of fatty acid with hormone-like actions-in the regulation of brain blood flow. The results will provide information on how to better use this technique to study brain function, which, in turn, may lead to a better understanding of certain illnesses and more effective treatments.

Healthy normal volunteers 18 years of age and older may be eligible for this study. Participants will fill out a health questionnaire and undergo a history, physical examination and MRI studies. MRI is a diagnostic tool that uses a strong magnetic field and radio waves instead of X-rays to show structural and chemical changes in tissues. During the scanning, the subject lies on a table in a narrow cylinder containing a magnetic field. An intercom system allows the subject to speak with the staff member performing the study at all times during the procedure. Four separate studies will be done-two carbon dioxide inhalation studies and two functional activation studies-as follows:

Carbon dioxide inhalation (indomethacin): This study is done in two parts. In both parts, an MRI brain scan is done. During the scan, the subject inhales an air mixture containing 6% carbon dioxide through a facemask or mouthpiece. Blood pressure and heart rate are monitored during inhalation of the mixture. For the second part of the study, indomethacin-a non-steroidal anti-inflammatory drug-is injected through a catheter (thin flexible tube) in an arm vein. Indomethacin inhibits prostaglandin production. Total scan time averages between 45 and 90 minutes, with a maximum of 2 hours.

Carbon dioxide inhalation (rofecoxib and celecoxib): This study is identical to the one above, except either rofecoxib or celecoxib is given instead of indomethacin. Both of these drugs are also non-steroidal anti-inflammatory drugs that inhibit prostaglandin production. Unlike indomethacin, rofecoxib and celecoxib are given orally instead of through a vein, so, to allow time for the drug to be absorbed, the second scan is delayed for 2 hours.

Functional activation (indomethacin): This study is done in two parts. In both parts, a MRI brain scan is done. During the study, the subject performs a simple motor task, such as finger tapping. For the second part of the study, indomethacin is injected through a catheter in an arm vein.

Functional activation (rofecoxib and celecoxib): This study is identical to the indomethacin functional activation study, except either rofecoxib or celecoxib is given instead of indomethacin. Because they are given orally instead of through a vein, the second scan is delayed 2 hours to allow time for the drug to be absorbed.

DETAILED DESCRIPTION:
Advances in MR perfusion imaging have provided clinical researchers with the opportunity to quantify regional increases in cerebral blood flow. The purpose of this study is to investigate in humans the role of prostaglandins in the regulation of cerebral blood flow during hypercapnia and functional activation. For this investigation the increase in cerebral blood flow associated with either hypercapnia or functional activation will be measured before and after the administration of pharmacological agents that inhibit the production of prostaglandins. In the hypercapnia study cerebral blood flow will be increased by inhalation of an air mixture containing 6% CO2. For the functional activation study cerebral blood flow will be increased by a sensory motor task.

ELIGIBILITY:
INCLUSION CRITERIA:

Any healthy normal volunteer above the age of 18 who is capable of giving informed consent.

EXCLUSION CRITERIA:

Subjects will be excluded for the following reasons.

They have contraindications to MR scanning, such as the following: aneurysm clip, implanted neural stimulator, implanted cardiac pacemaker or autodefibrillator, cochlear implant, ocular foreign body (e.g., metal shavings), or insulin pump.

They have panic disorder or migraine (because of possible complications with CO2 inhalation).

They have cirrhosis, any renal dysfunction, or a chronic respiratory illness (such as asthma).

They have allergies to sulfonamide drugs or cyclo-oxygenase inhibitors (NSAIDS).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 125
Dates: Start 2000-09; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] O'Banion MK. Cyclooxygenase-2: molecular biology, pharmacology, and neurobiology. Crit Rev Neurobiol. 1999;13(1):45-82. doi: 10.1615/critrevneurobiol.v13.i1.30. PMID 10223523
- [Background] Kaufmann WE, Worley PF, Pegg J, Bremer M, Isakson P. COX-2, a synaptically induced enzyme, is expressed by excitatory neurons at postsynaptic sites in rat cerebral cortex. Proc Natl Acad Sci U S A. 1996 Mar 19;93(6):2317-21. doi: 10.1073/pnas.93.6.2317. PMID 8637870
- [Background] Yamagata K, Andreasson KI, Kaufmann WE, Barnes CA, Worley PF. Expression of a mitogen-inducible cyclooxygenase in brain neurons: regulation by synaptic activity and glucocorticoids. Neuron. 1993 Aug;11(2):371-86. doi: 10.1016/0896-6273(93)90192-t. PMID 8352945